CLINICAL TRIAL: NCT01837069
Title: Optimization of Pre-surgical Testing With an Intensive Multifactorial Intervention to MinimiZe Cardiovascular Events in Orthopedic Surgery
Brief Title: Risk Factor Control Before Orthopedic Surgery
Acronym: OPTMIZE-OS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment / DSMB approval to halt recruitment
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-02407
Record Dates: First submitted 2013-04-12; First posted 2013-04-22 (Estimated); Results first posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Osteoarthritis; Cardiovascular Disease
Keywords: Hypertension; Diabetes; Coronary Artery Disease; Peripheral Vascular Disease
MeSH Terms: conditions — Osteoarthritis; Cardiovascular Diseases; Hypertension; Diabetes Mellitus; Coronary Artery Disease; Peripheral Vascular Diseases | interventions — Metoprolol; Adrenergic beta-Antagonists; Lisinopril; Angiotensin-Converting Enzyme Inhibitors; Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): Lifestyle counseling (nutrition, physical activity, medication compliance and smoking cessation) Atorvastatin 80mg PO QD Metoprolol 25mg PO BID if HR is elevated Lisinopril 2.5 mg PO QD if SBP is elevated
  Interventions: Drug: Metoprolol; Drug: Lisinopril; Drug: Atorvastatin; Behavioral: Lifestyle counseling
- Control (No Intervention): Standard of care

INTERVENTIONS:
Drug: Metoprolol — 25mg PO BID if the HR is elevated at preadmission testing
  Other Names: Beta blocker
  Arms: Treatment
Drug: Lisinopril — 2.5mg PO QD if the HR is elevated at preadmission testing
  Other Names: ACE inhibitor
  Arms: Treatment
Drug: Atorvastatin — 80mg PO QD at preadmission testing
  Other Names: Statin
  Arms: Treatment
Behavioral: Lifestyle counseling — Diet, exercise, medication adherance and smoking counseling
  Arms: Treatment

SUMMARY:
This trial is designed to determine the best preoperative management strategy for patients undergoing orthopedic surgery.

DETAILED DESCRIPTION:
OPTIMIZE - OS (Optimization of Pre-surgical Testing with an Intensive Multifactorial Intervention to MinimiZe Cardiovascular Events - Orthopedic Surgery) trial is to determine the best management strategy for patients undergoing orthopedic surgery. OPTIMIZE will be a prospective randomized trial that will enroll patients during pre-surgical testing before orthopedic surgery. This trial will investigate different strategies aimed at lowering cardiovascular events following orthopedic surgery. The study will compare an intensive multifactorial intervention comprising behavioral modification and polypharmacologic therapy aimed at several modifiable risk factors versus usual care. The trial hypothesis is that a personalized optimization approach is superior to usual care in reducing a composite of death, myocardial infarction, stroke, transient ischemic attack, myocardial necrosis, venous thromboembolism or thrombosis requiring reoperation at 30-days. Secondary endpoints include length of stay, major bleeding, each individual endpoint from the primary endpoint, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* • ≥ 21 years of age

  * Subjects undergoing open orthopedic surgery of the hip, knee or spine
  * Surgery is scheduled at least 3 days after PAT visit and no more than 14 days.
  * High risk subject cohort

    * Coronary artery disease, or
    * Cerebrovascular disease (prior stroke, TIA or carotid artery disease (>70% stenosis), or
    * Peripheral artery disease, or
    * Prior Venous thromboembolism or arterial thromboembolism, or
    * Age ≥ 60 years and 2 of the following
  * Renal insufficiency (creatinine clearance < 60ml/min)
  * Diabetes
  * COPD
  * Hypertension
  * Active smoker or stopped less than 30 days prior to consent
  * Cancer (excluding BCC)
  * Heart Failure

Exclusion Criteria:

* • Known intolerance to statins

  * Subject is already on maximum dose statin (atorvastatin/Lipitor 80mg daily or rosuvastatin/crestor 40mg daily)
  * Bilateral renal artery stenosis
  * End stage renal disease (receiving dialysis or CrCl <30ml/min)
  * Known allergy or intolerance to ACE-inhibitor (other than cough) or Angiotensin receptor blocker (e.g. angioedema, hyperkalemia)
  * Known allergy or intolerance to beta blockers
  * Known sick sinus syndrome not treated with permanent pacemaker
  * Known greater than first degree AV block not treated with a pacemaker
  * Excessive alcohol intake
  * Acute Coronary Syndrome requiring hospitalization within 1 month
  * Stroke within 1 month
  * Known pregnancy
  * Severe co-morbid condition with life expectancy < 6 months
  * Inability to give informed consent or adhere to follow-up as per protocol
  * Current participation in another investigational drug or device trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2014-02; Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Berger, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Hospital for Joint Diseases, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 103 | 95
Completed | 103 | 95
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 103 | 95 | 198
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 103 | 95 | 198
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 44 | 100
  Male | 47 | 51 | 98
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 3 | 6
  Black or African American | 14 | 12 | 26
  White | 80 | 74 | 154
  Hispanic or Latino | 10 | 11 | 21
  # Unknown or not reported | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 103 | 95 | 198

OUTCOME MEASURES:

1. Primary Outcome: Number of Partipants That Experienced Death, Myocardial Infarction, Stroke, Transient Ischemic Attack, Myocardial Necrosis, or Venous Thromboembolism
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 103 | 95
participants | 10 | 2

2. Secondary Outcome: Modified Composite of Cardiovascular Events
Description: the reduction in the composite of death, myocardial infarction, stroke, transient ischemic attack, myocardial necrosis, venous thromboembolism, or reoperation
Time Frame: 30 days
Population: No data are available for this Outcome Measure. Multiple efforts were made to obtain the data from the PI but were unsuccessful, therefore, data cannot be reported.
Arm/Group | Treatment | Control
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Length of Stay
Time Frame: Hospital stay, ~7 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Treatment | Control
Number analyzed (Participants) | 93 | 89
days | 3 [2 to 4] | 3 [2 to 3.75]

4. Other Pre Specified Outcome: Each Individual Endpoint of the Composite of Cardiovascular Events
Time Frame: 30 days
Population: Efforts were made to collect this data from PI, but data analysis was not completed for this outcome measure
Arm/Group | Treatment | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/95
Other Adverse Events (participants affected / at risk) | 0/103 | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT01837069/Prot_SAP_000.pdf